CLINICAL TRIAL: NCT02760095
Title: Effects of Environmental Enteric Dysfunction (EED) on Zinc (Zn) Absorption and Retention in Young Children: Study 1 - Absorption of Zn and Vitamin A From a Standard Dose
Brief Title: Effects of EED on Zn Absorption and Retention in Children From a Standard Dose
Acronym: ZEED1
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Other Study IDs: 14-2430A
Record Dates: First submitted 2015-07-24; First posted 2016-05-03 (Estimated); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Environmental Enteric Dysfunction; Zinc Deficiency; Vitamin A Deficiency
Keywords: environmental enteric dysfunction; environmental enteropathy; zinc; vitamin A; Bangladesh
MeSH Terms: conditions — Vitamin A Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Spot urine samples x 4 days; complete fecal collections x 4 days; blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Children with EED: Children are placed in this arm if they screen positive for EED using the urinary lactulose:mannitol (L:M) recovery ratio. Children will receive a one-time 3 mg standard dose of zinc sulfate with stable isotope zinc tracer and 0.5 mg standard dose of 13C10-retinyl-acetate (vitamin A isotope).
  Interventions: Drug: 3 mg zinc sulfate supplement; Drug: 0.5 mg of 13C10-retinyl-acetate
- Children without EED: Children are placed in this arm if they screen negative for EED using the urinary lactulose:mannitol (L:M) recovery ratio. Children will receive a one-time 3 mg standard dose of zinc sulfate with stable isotope zinc tracer and 0.5 mg standard dose of 13C10-retinyl-acetate (vitamin A isotope).
  Interventions: Drug: 3 mg zinc sulfate supplement; Drug: 0.5 mg of 13C10-retinyl-acetate

INTERVENTIONS:
Drug: 3 mg zinc sulfate supplement
Drug: 0.5 mg of 13C10-retinyl-acetate
  Other Names: Vitamin A isotope

SUMMARY:
The overall objective is to determine the impact of EED on zinc absorption and homeostasis, and its impact on the absorptive capacity of vitamin A absorption of young children (18-24 months of age) in an austere setting with high rates of diarrhea, stunting, and micro-nutrient deficiencies.

DETAILED DESCRIPTION:
Participating children are screened for EED using the lactulose:mannitol ratio test and assigned to one of two groups: +EED or -EED. All participants will be given standard, physiological dose of 3 mg zinc sulfate with a zinc stable isotope tracer on study day 8.

On study day 11, 0.5 mg of 13C10-retinyl-acetate will be administered orally to all participants.

Spot urine samples will be collected twice daily from study days 11-14. Complete fecal collections will be obtained for days 11-14. Duplicate diets of all foods consumed will be collected on days 11-14. On study day 14, a blood sample will be taken for analysis of vitamin A isotope status.

ELIGIBILITY:
Inclusion Criteria:

* Absence of apparent health problems that would impair ability to consume regular diet, to tolerate zinc supplements, or to comply with demands of metabolic studies
* Length for age Z-score (LAZ) between -1.5 to -3.0
* Hemoglobin (Hgb) ≥ 8

Exclusion Criteria:

* Outside age range
* Hgb < 8
* Chronic illness
* Recent diarrhea (within past 2 weeks, treated with supplemental zinc)
* Severe stunting and/or severe acute malnutrition (SAM): LAZ <-3; Weight-for-age Z-score (WHZ) <-3 or mid-upper arm circumference (MUAC) < 115 or edema

Ages: 18 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Toddlers aged 18-24 mos living in Dhaka, Bangladesh
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Absorption of zinc (AZ) from standard dose | 1 day
  Absorption of zinc from standard 3 mg dose will be measured using zinc isotope tracer methods
Endogenous fecal zinc (EFZ) | 4 days
  EFZ measured from zinc isotope ratios in complete fecal collections
Vitamin A absorption | 1 day
  Absorption efficiency of retinol will be measured by isotope ratios in blood

SECONDARY OUTCOMES:
Plasma zinc | 1 day
  Plasma zinc concentration
Alkaline phosphatase | 1 day
Serum retinol | 1 day
Methyl malonic acid | 1 day
  serum
Vitamin B12 | 1 day
Serum ferritin | 1 day
Soluble transferrin receptors | 1 day
C-reactive Protein (CRP) | 1 day
Alpha-Glycoprotein (AGP) | 1 day
Tumor necrosis factor (TNF) alpha | 1 day
Serum endocab | 1 day
Fecal neopterin | 1 day
Myeloperoxidase | 1 day
Alpha 1 antitrypsin | 1 day
Calprotectin | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Nancy F Krebs, MD, MS, Principal Investigator — University of Colorado, Denver
Locations (2):
- University of Colorado Denver School of Medicine, Aurora, Colorado, United States
- icddr,b (International Centre for Diarrheal Disease Research, Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mondal P, Long JM, Westcott JE, Islam MM, Ahmed M, Mahfuz M, Ahmed T, Miller LV, Krebs NF. Zinc Absorption and Endogenous Fecal Zinc Losses in Bangladeshi Toddlers at Risk for Environmental Enteric Dysfunction. J Pediatr Gastroenterol Nutr. 2019 Jun;68(6):874-879. doi: 10.1097/MPG.0000000000002361. PMID 31033623